CLINICAL TRIAL: NCT03271801
Title: Skills Training in Stimulus Control of Meals and Snacks Within a Family-based Obesity Treatment Intervention
Brief Title: Skills Training Within a Family-based Obesity Treatment Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment Challenges
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Shannon Robson, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 906996-1
Record Dates: First submitted 2017-03-29; First posted 2017-09-05 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child Health Education (Active Comparator): The child health education condition will participate in a family-based obesity treatment program for the first 40 minutes of each session, followed by 20 minutes designated to education about a child health topic. Parents and children will be asked to self-monitor sugar-sweetened beverages, fruits, vegetables, and minutes of physical activity and screen time.
  Interventions: Behavioral: child health education
- Skills Training (Experimental): The skills training condition will participate in a family-based obesity treatment program for the first 40 minutes of each session followed by 20 minutes of experiential learning about meal stimulus control strategies. Parents and children will be asked to self-monitor sugar-sweetened beverages, fruits, vegetables, and minutes of physical activity and screen time. In addition they will self-monitor the use the following stimulus control strategies: portion control, energy density and variety.
  Interventions: Behavioral: skills training

INTERVENTIONS:
Behavioral: child health education — 10, 60-minute sessions with a family-based obesity treatment program implemented for the first 40-minutes of each session followed by 20 minutes of education about a child health topic.
  Arms: Child Health Education
Behavioral: skills training — 10, 60-minute sessions with a family-based obesity treatment program implemented for the first 40-minutes of each session followed by 20 minutes of experiential learning about stimulus control strategies (portion size, energy density, variety).
  Arms: Skills Training

SUMMARY:
This study is investigating the impact of a skills training program in stimulus control of meals and snacks on zBMI. Participants will be randomized to a standard family-based obesity treatment intervention with education on child health or a standard family-based obesity treatment intervention with experiential learning about meal stimulus control strategies.

DETAILED DESCRIPTION:
Family-based obesity treatment interventions can successfully reduce weight in children, but are often limited in the practice of skills being taught during treatment sessions.

Skills training focused on a particular behavioral strategy can provide parents with an experiential component of learning where the information learned as part of a family-based obesity treatment intervention is also practiced. Health education simply provides knowledge to a family about a topic.

ELIGIBILITY:
Inclusion Criteria:

* caregiver of child is ≥18 years of age;
* the caregiver has a child between the ages of 4 and 8 years-old who is classified as overweight (body mass index for age ≥ 85th percentile);
* the caregiver and child are able to read, speak and understand English due to delivery of the program in English;
* has transportation to the University of Delaware; and
* is willing and able to commit to the 3-month study.

Exclusion Criteria:

* the child has a medical condition impacting physical activity or eating (e.g. Type

  1 or Type 2 diabetes);
* the child have a medical condition that affects growth (e.g. Prader Willi Syndrome);
* the child is currently participating in a weight management program, and/or taking weight loss medication; or
* the caregiver or child has an inability to participate in regular physical activity.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
z-BMI | 3-months
  Height and weight will be used to calculate BMI (kg/m2) and BMI will be standardized in relation to the population mean and standard deviation for the child's age to sex to determine zBMI.

SECONDARY OUTCOMES:
Energy intake | 3-months
  Based upon a 3-day dietary record analyzed using NDS-R, energy intake will be averaged across the three days.
Percent Energy from Fat | 3-months
  Based upon a 3-day dietary record analyzed using NDS-R, the calories from fat will be divided by total energy intake (calories) to get percentage energy from fat.
Food groups servings | 3-months
  Based upon a 3-day dietary record analyzed using NDS-R, the number of servings consumed from each food group will be averaged over three days.
Physical Activity | 3-months
  Minutes spent engaging in moderate-to-vigorous physical activity will be measured using the PD-PAR.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Robson, PhD, MPH, RD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No